CLINICAL TRIAL: NCT04280549
Title: Platelet PAR-1 Activation in Health and Diabetes
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Joshua Beckman, Professor, Vanderbilt University Medical Center
Other Study IDs: 192207
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Subjects: Subjects will have a single visit where a short medical history/list of current medications and single blood draw will be performed.
- Type 2 Diabetic Subjects: Subjects will have a single visit where a short medical history/list of current medications and single blood draw will be performed.

SUMMARY:
Platelet activation has been associated with bad events like heart attack and stroke. There are a variety of platelet activators that regulate how active a platelet is. We are interested in Protease-activated receptors (PAR)-1. We are currently studying PAR-1 activation in persons with severe peripheral artery disease. We seek, through this project, to understand PAR-1 activation in persons without peripheral artery disease. As many patients with peripheral artery disease have diabetes, we will also evaluate PAR-1 activation in persons with type 2 diabetes. In addition we will assess the impact of the glucagon-like peptide (GLP)-1 signaling pathway on platelet activation. Levels of platelet activation will be determined using platelet aggregation experiments and assessment of platelet-monocyte aggregates in peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women ≥60 years of age OR
* Type 2 diabetic men and women ≥60 years of age

Exclusion Criteria:

* Active cancer
* Prior myocardial infarction, prior stroke, diagnosed peripheral artery disease
* Severe liver (cirrhosis, cancer, or end-stage liver disease), kidney disease (eGFR <30 cc/min).
* Pregnancy or lactation
* Active vasculitis
* Anticipated lifespan < 2 years
* Current use of a DOAC

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic and healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Platelet Activation | One day
  Number of dilysyl-MDA cross-links formed in human platelets
Protease Activated Receptor-1 Activation | One day
  Number of cleaved PAR-1 receptors in proportion to number of uncleared PAR-1 receptors

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Beckman, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. (Link to be provided).